CLINICAL TRIAL: NCT00510328
Title: Vibration Therapy Effects on Muscle Firing Patterns
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD0607060023
Record Dates: First submitted 2007-07-31; First posted 2007-08-02 (Estimated); Last update posted 2007-08-02 (Estimated); Status verified 2007-07

CONDITIONS: Healthy
Keywords: whole body vibration; muscle physiology

INTERVENTIONS:
Device: Whole Body Vibration

SUMMARY:
The purpose of this study is to determine the effects of whole body vibration therapy on muscle firing patterns as measured by EMG analysis.

DETAILED DESCRIPTION:
Proprioception is the specialized sensory modality that informs the body as to movement, position, and spatial orientation through mechanisms that track sensations accompanying joint movement and position. Mechanoreceptors in joints, along with vestibular, visual, muscle spindle, Golgi tendon organ, ligament and tendon sensory receptors, comprise the propriosensory system, which conveys information to the motor system to maintain equilibrium on a reflexive, automatic basis. Alterations in somatosensory input from mechanoreceptors have been identified as causing aberrant muscle firing patterns.

ELIGIBILITY:
Inclusion Criteria:

* Logan student, staff, or faculty with no history of ankle injury
* Ages 18 - 60 years old
* Logan student, staff, or faculty with no history of ankle surgery
* No visual or vestibular condition that would affect balance

Exclusion Criteria:

* Systemic illnesses that have an adverse effect on balance
* Local infection, injury, or other malignancy affecting the lower extremity
* Any unstable joints of the lower extremity
* Any spinal manipulation within 48 hours
* Prescription or herbal muscle stimulants, relaxants, etc. that could affect balance
* Pregnancy

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Electromyographic analysis of the gastrocnemius muscle

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E. Enix, DC, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan University, College of Chiropractic, Chesterfield, Missouri, United States